CLINICAL TRIAL: NCT03394989
Title: A Multicenter, Randomized, Parallel-group, Placebo-controlled, 4-week Clinical Endpoint Bioequivalence Study Comparing Fluticasone Propionate/Salmeterol 100/50 µg Inhalation Powder With Advair® Diskus 100/50 µg in Asthma Patients
Brief Title: BE Study of Fluticasone Propionate/Salmeterol Inhalation Powder in Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cipla Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U-FS-MU-AS3120
Record Dates: First submitted 2017-12-26; First posted 2018-01-09 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2019-11

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, parallel-group, placebo-controlled
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test (Experimental): Fluticasone propionate/salmeterol 100/50 µg
  Interventions: Drug: Fluticasone propionate/salmeterol 100/50 µg
- Comparator (Active Comparator): Fluticasone propionate/salmeterol 100/50 µg
  Interventions: Drug: Advair Diskus 100/50 Dry Powder Inhaler, 60 ACTUAT
- Placebo (Other): Test Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol 100/50 µg — Test Arm: Dry powder inhaler
  Arms: Test
Other: Placebo — Placebo
  Arms: Placebo
Drug: Advair Diskus 100/50 Dry Powder Inhaler, 60 ACTUAT — Comparator Arm: Dry powder inhaler
  Arms: Comparator

SUMMARY:
The purpose of this study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product in adult patients with asthma.

DETAILED DESCRIPTION:
This study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product in terms of FEV1 measured at different time-points in adult patients with asthma.

ELIGIBILITY:
Inclusion Criteria

1. Patients who have signed informed consent form before initiation of any study related procedure.
2. Male or female patients who are ≥18 years of age at the time informed consent is obtained.
3. Documented diagnosis of asthma as defined by the National Asthma Education and Prevention Program (NAEPP) and diagnosed at least 12 weeks prior to screening.
4. Patients with pre-bronchodilator forced expiratory volume in one second (FEV1) of 40% to 85% (both inclusive) of the predicted normal value at the Screening Visit V2.
5. Patients who demonstrated an increase of ≥15% of FEV1 within 15 30 minutes following administration of albuterol at Screening Visit V2
6. Patients who are stable on current asthma treatment for at least 4 weeks prior to Screening Visit V1.
7. Patients who are able to discontinue their current asthma medications (if any) and any other prohibited medications throughout the study, per the protocol list of prohibited medications during study participation (see Section 6.3.2).
8. Patients who are able to replace their current short-acting beta 2 agonist (SABA) inhaler with the study provided albuterol inhaler to be used as rescue medicine (as needed) throughout the study. Patients who are able to withhold SABAs for at least 6 hours prior to lung function assessments on study visits.
9. Patient who are non-smokers or ex-smokers; and have had ≤10 pack years
10. Patients who have not inhaled tobacco or consumed other tobacco containing products have not inhaled vaping products, drugs of abuse, or inhaled marijuana for at least 12 months prior to screening.
11. Women of childbearing potential (WOCBP) must not be lactating or pregnant at screening, as documented by a negative screening pregnancy test
12. Women of childbearing potential must commit to consistent and correct use of an acceptable method of birth control (at the investigator's discretion) throughout the study.

Exclusion criteria:

1. History of life-threatening asthma defined as an asthma episode(s) that required intubation and/or was associated with hypercapnic, respiratory arrest, or hypoxic seizures, asthma related syncopal episode(s) within the past one year.
2. History of any asthma-related hospitalizations within the past one year.
3. Any asthma exacerbation requiring emergency room (ER) visits or systemic (including oral) corticosteroids within 2 months prior to signing the consent.
4. Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia (prolonged QT interval as judged by the investigator). In addition, historical or current evidence of significant hematologic, hepatic neurologic, psychiatric, renal, or other diseases that in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
5. Patients with uncontrolled allergic rhinitis.
6. Clinical visual evidence of oral candidiasis.
7. History of any adverse reaction; known hypersensitivity to any sympathomimetic drug
8. Use of medication(s) with potential to affect the course of asthma or to interact with sympathomimetic amines throughout the study period.
9. Recent viral or bacterial infection or infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 4 weeks of screening.
10. Patients, who in the opinion of the investigator, significantly abuse alcohol or drugs will be excluded.
11. Use of systemic (including oral) corticosteroids within 4 weeks or intramuscular depot corticosteroid treatment 90 days prior to screening for any reason other than asthma (see exclusion criteria #3 above).
12. Patients taking any immunosuppressive medications within 4 weeks prior to screening and during the study.
13. Factors (e.g., infirmity, disability, geographic location) that the investigator felt would likely limit the patients' compliance with the study protocol or scheduled clinic visits.
14. Use of any investigational drug (approved or unapproved) within 30 days
15. Study participation by clinical investigator site employees and/or their immediate relatives.
16. Patients who are unable to produce valid and reproducible spirometry per American Thoracic Society/European Respiratory Society (ATS/ERS) standards at the screening visit or unable to use the electronic diary (e diary).
17. Patients unable to use the inhalation powder device adequately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1366 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Area under the serial Force Expiration volume1 from time 0 to 12 hours (AUC0-12 hours) | one day
  Area under the serial Force Expiration volume1 from time 0 to 12 hours (AUC0-12 hours) on the first day of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Research Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No